CLINICAL TRIAL: NCT05381558
Title: Evaluation of the Role of Local Steroid Injection in Treatment of Idiopathic Spasmodic Flat Foot in Adolescent Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Pemen Phillip Adely, resident doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Spasmodic faltfoot
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Flatfoot
MeSH Terms: conditions — Flatfoot | interventions — Triamcinolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- spasmotic flatfoot patient (Experimental)
  Interventions: Drug: Triamcinolone Injection

INTERVENTIONS:
Drug: Triamcinolone Injection — local injection in sinus tarsi

SUMMARY:
* Population: adolescent patients aged from 10 to 16 years
* Interventions:

  1. Examination under general anaesthesia if the deformity corrected spontaneously
  2. local injection of steroid in sinus tarsi
  3. cast in varus for 6 weeks
* Outcomes: primary outcome : Evaluate the clinical and functional outcomes according AOFAS.
* Time: follow up within one and half month, 3 months, 6 months, one year.

DETAILED DESCRIPTION:
• Does local steroid injection have a role in treatment of spasmodic flat foot in adolescent patients? One of the most common foot complaints in the juvenile and adolescent age group is the "flatfoot" deformity. (1) Clinical evaluation of flatfeet primarily focuses on differentiation between the two main types: flexible and rigid. (2) The flexible type is a common diagnosis and is one which is usually not problematic and rarely needs treatment. (3) Rigid flatfoot deformity is less common (occurring one-third as often as the flexible type) but often is symptomatic and requires treatment. (4) Spasmodic valgus foot is usually associated with resistant pain and deformity. It shows controversy regarding its incidence, etiology, and treatment. (5) Spasmodic flatfoot is a rare condition characterized by a rigid and usually painful valgus deformity in the hind foot with peroneal muscles spasms (6,7) It is often caused by inter-tarsal bars or bone anomalies that restrict tarsal joint motion . (8) Our study aims to evaluate the functional and clinical outcome after local long-acting steroid injection in the sinus tarsi followed by cast in adolescent patients with spasmodic flatfeet without coalition.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patients from 10 to 16 years
* Flat foot with peroneal muscle spasm

Exclusion Criteria:

* Flatfoot uncorrected by manipulation under general anaesthesia

  * neuromuscular disorders
  * evidence of coalition in CT or MRI

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the functional outcomes according AOFAS Ankle-hindfoot scale | 45days

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] BLOCKEY NJ. Peroneal spastic flat foot. J Bone Joint Surg Br. 1955 May;37-B(2):191-202. doi: 10.1302/0301-620X.37B2.191. No abstract available. PMID 14381462
- [Background] Jayakumar S, Cowell HR. Rigid flatfoot. Clin Orthop Relat Res. 1977 Jan-Feb;(122):77-84. PMID 837623
- [Background] Harris EJ, Vanore JV, Thomas JL, Kravitz SR, Mendelson SA, Mendicino RW, Silvani SH, Gassen SC; Clinical Practice Guideline Pediatric Flatfoot Panel of the American College of Foot and Ankle Surgeons. Diagnosis and treatment of pediatric flatfoot. J Foot Ankle Surg. 2004 Nov-Dec;43(6):341-73. doi: 10.1053/j.jfas.2004.09.013. No abstract available. PMID 15605048
- [Background] Luhmann SJ, Rich MM, Schoenecker PL. Painful idiopathic rigid flatfoot in children and adolescents. Foot Ankle Int. 2000 Jan;21(1):59-66. doi: 10.1177/107110070002100111. PMID 10710264
- [Background] HARRIS RI, BEATH T. Etiology of peroneal spastic flat foot. J Bone Joint Surg Br. 1948 Nov;30B(4):624-34. No abstract available. PMID 18894612